CLINICAL TRIAL: NCT00292032
Title: Cardiac Arrest Survivors With Preserved Ejection Fraction Registry (CASPER)
Brief Title: Registry of Unexplained Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Kingston Health Sciences Centre (Other); Quebec Heart Institute (Other); The Queen Elizabeth Hospital (Other); St. Boniface Hospital (Other); Unity Health Toronto (Other); Vancouver Island Health Authority (Other); Provincial Health Services Authority British Columbia (Other); Montreal Heart Institute (Other); Ottawa Heart Institute Research Corporation (Other); University of Calgary (Other)
Responsible Party: Principal Investigator, Andrew Krahn, Principal Iinvestigator, University of British Columbia
Other Study IDs: R-04-099; 10076 (Other: REB)
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Cardiac Arrest; Long QT Syndrome; Brugada Syndrome; Catecholaminergi Polymorphic Ventricular Tachycardia; Idiopathic VentricularFibrillation; Early Repolarization Syndrome; Arrhythmogenic Right Ventricular Cardiomyopathy
Keywords: cardiac arrest; diagnosis; genetics; testing
MeSH Terms: conditions — Heart Arrest; Long QT Syndrome; Brugada Syndrome; Arrhythmogenic Right Ventricular Dysplasia; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cardiac Arrest Survivors or Post Mortem Unexplained Cardiac: Probands - Unexplained Cardiac Arrest Survivors and Post Mortem Unexplained Cardiac Arrest Cases
- First Degree Family Members: First Degree Family Members of those affected by Sudden Unexplained Cardiac Arrest

SUMMARY:
The CASPER will collect systematic clinical assessments of patients and families within the multicenter Canadian Inherited Heart Rhythm Research Network. Unexplained Cardiac Arrest patients and family members will undergo standardized testing for evidence of primary electrical disease and latent cardiomyopathy along with clinical genetics screening of affected individuals based on an evident or unmasked phenotype.

DETAILED DESCRIPTION:
Arrhythmias caused by congenital or acquired abnormalities of cardiac K+ or Na+ channels are increasingly recognized as a cause of syncope and sudden death. Cardiac arrest in the absence of overt structural heart disease was previously considered idiopathic ventricular fibrillation (IVF). The list of causes of "unexplained" cardiac arrest (UCA) now encompasses K+ related abnormalities (Long and Short QT, Andersen's), Na+ related (Long QT3, Brugada), Ca++ related (Catecholaminergic Polymorphic Ventricular Tachycardia-CPVT), and latent cardiomyopathy. These underlying causes of cardiac arrest are overtly familial in 30-60% of cases. Clinical detection of the underlying phenotype is crucial to direct appropriate treatment, genetic testing and screening of family members.

Phenotype recognition of the range of these rare genetic conditions includes non-invasive and invasive testing to demonstrate the hallmarks of each individual condition, and exclude common causes such as ischemic or idiopathic forms of cardiomyopathy. The outcomes from this type of testing have not been assessed in a systematic fashion in patients with UCA or their family members. Phenotype-genotype correlation is necessary to develop optimal diagnostic testing in probands and screening techniques in their family members, which will result in disease-specific therapy. Genetic testing of patients with an overt phenotype demonstrates a potentially causative mutation in 50-75% of LQTS patients, and 20% of Brugada's Syndrome patients. Despite recognized mutations with phenotypic expression models, 30-80% of patients will have negative gene screening despite overt or latent clinical disease.

The proposed project is evaluating a systematic approach to clinical assessment and genetic screening of patients and families with UCA and suspected inherited arrhythmias involving:

1. A multicenter registry of UCA patients, their family members and referred patients with familial sudden death undergoing standardized testing for evidence of primary electrical disease (PED). The single center pilot experience at the applicant's institution has proven feasibility, and has been accepted for publication in Circulation, indicating novelty. Ten centers across Canada have agreed to participate. The target is to enroll 1500 UCA probands, 1st degree family members. 1st degree relatives of autopsy negative unexplained sudden death victims.
2. Long term cardiac monitoring for (3 years) in select high-risk patients with an injectable cardiac monitor to detect potential substrate and/ore triggers for sudden death.
3. DNA/plasma collection and biobanking for stratified whole exome sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrest requiring cardioversion or defibrillation.
* Syncope with documented polymorphic ventricular tachycardia felt to be responsible for the index event.
* First degree relative of an index case of UCA undergoing clinical testing.
* First degree relative of a family member with UCA or sudden death before age 35 with a negative autopsy for cause of death, presumed arrhythmic.
* First degree relative of a family member with UCA or sudden death with objective evidence of primary electrical disease, such as a diagnostic electrocardiogram (ECG), exercise test, drug infusion, or genetic testing.

Exclusion Criteria:

* Coronary artery disease (stenosis > 50%)
* Reduced left ventricular function (left ventricular ejection fraction [LVEF] < 50%)
* Event managed without an implantable cardioverter defibrillator [ICD] (for follow-up portion)
* Unwilling or unable to provide clinical follow-up (for follow-up portion)
* Comorbidity making survival of > 1 year unlikely
* Persistent resting QTc > 460 msec for males and 480 msec for females
* Reversible cause of cardiac arrest such as marked hypokalemia (< 2.8 mmol/l) or drug overdose sufficient in gravity without other cause to explain the cardiac arrest
* Hemodynamically stable sustained monomorphic ventricular tachycardia with a QRS morphology consistent with recognized forms of idiopathic ventricular tachycardia (outflow tract or apical septal)
* Brugada's sign with e2 mm ST elevation in V1 and/or V2
* Unwilling or unable to provide consent

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Unexplained cardiac arrest patients, and first degree relatives of 1) UCA patients 2) patients with known primary electrical disease or 3) unexplained sudden death before age 60
Sampling Method: Non-Probability Sample
Enrollment: 1529 (Actual)
Dates: Start 2004-05; Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Developing and Testing Algorithms for Diagnostics and Treatments in Survivors of Unexplained Cardiac Arrest | 25 years
  Long Term follow up data on survivors of cardiac arrest Long term monitoring of high risk patients and familymembers with an Injectable Cardiac Monitor 24 hour holter monitoring during provocative testing with epinephrine infusion and ambulatory activities to detect subclinical repolarization

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Krahn, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Krahn AD, Gollob M, Yee R, Gula LJ, Skanes AC, Walker BD, Klein GJ. Diagnosis of unexplained cardiac arrest: role of adrenaline and procainamide infusion. Circulation. 2005 Oct 11;112(15):2228-34. doi: 10.1161/CIRCULATIONAHA.105.552166. Epub 2005 Oct 3. PMID 16203906
- [Result] Krahn AD, Healey JS, Chauhan V, Birnie DH, Simpson CS, Champagne J, Gardner M, Sanatani S, Exner DV, Klein GJ, Yee R, Skanes AC, Gula LJ, Gollob MH. Systematic assessment of patients with unexplained cardiac arrest: Cardiac Arrest Survivors With Preserved Ejection Fraction Registry (CASPER). Circulation. 2009 Jul 28;120(4):278-85. doi: 10.1161/CIRCULATIONAHA.109.853143. Epub 2009 Jul 13. PMID 19597050
- [Derived] Davies B, Bartels K, Hathaway J, Xu F, Roberts JD, Tadros R, Green MS, Healey JS, Simpson CS, Sanatani S, Steinberg C, Gardner M, Angaran P, Talajic M, Hamilton R, Arbour L, Seifer C, Fournier A, Joza J, Krahn AD, Lehman A, Laksman ZWM. Variant Reinterpretation in Survivors of Cardiac Arrest With Preserved Ejection Fraction (the Cardiac Arrest Survivors With Preserved Ejection Fraction Registry) by Clinicians and Clinical Commercial Laboratories. Circ Genom Precis Med. 2021 Jun;14(3):e003235. doi: 10.1161/CIRCGEN.120.003235. Epub 2021 May 7. PMID 33960826
- [Derived] Cheung CC, Davies B, Gibbs K, Laksman ZW, Krahn AD. Patch monitors for arrhythmia monitoring in patients for suspected inherited arrhythmia syndrome. J Cardiovasc Electrophysiol. 2021 Mar;32(3):856-859. doi: 10.1111/jce.14917. Epub 2021 Feb 15. PMID 33512057
- [Derived] Mellor G, Laksman ZWM, Tadros R, Roberts JD, Gerull B, Simpson CS, Klein GJ, Champagne J, Talajic M, Gardner M, Steinberg C, Arbour L, Birnie DH, Angaran P, Leather R, Sanatani S, Chauhan VS, Seifer C, Healey JS, Krahn AD. Genetic Testing in the Evaluation of Unexplained Cardiac Arrest: From the CASPER (Cardiac Arrest Survivors With Preserved Ejection Fraction Registry). Circ Cardiovasc Genet. 2017 Jun;10(3):e001686. doi: 10.1161/CIRCGENETICS.116.001686. PMID 28600387
- [Derived] Steinberg C, Padfield GJ, Champagne J, Sanatani S, Angaran P, Andrade JG, Roberts JD, Healey JS, Chauhan VS, Birnie DH, Janzen M, Gerull B, Klein GJ, Leather R, Simpson CS, Seifer C, Talajic M, Gardner M, Krahn AD. Cardiac Abnormalities in First-Degree Relatives of Unexplained Cardiac Arrest Victims: A Report From the Cardiac Arrest Survivors With Preserved Ejection Fraction Registry. Circ Arrhythm Electrophysiol. 2016 Sep;9(9):e004274. doi: 10.1161/CIRCEP.115.004274. PMID 27635072
- [Derived] Herman AR, Cheung C, Gerull B, Simpson CS, Birnie DH, Klein GJ, Champagne J, Healey JS, Gibbs K, Talajic M, Gardner M, Bennett MT, Steinberg C, Janzen M, Gollob MH, Angaran P, Yee R, Leather R, Chakrabarti S, Sanatani S, Chauhan VS, Krahn AD. Outcome of Apparently Unexplained Cardiac Arrest: Results From Investigation and Follow-Up of the Prospective Cardiac Arrest Survivors With Preserved Ejection Fraction Registry. Circ Arrhythm Electrophysiol. 2016 Jan;9(1):e003619. doi: 10.1161/CIRCEP.115.003619. PMID 26783233
- [Derived] Krahn AD, Healey JS, Chauhan VS, Birnie DH, Champagne J, Sanatani S, Ahmad K, Ballantyne E, Gerull B, Yee R, Skanes AC, Gula LJ, Leong-Sit P, Klein GJ, Gollob MH, Simpson CS, Talajic M, Gardner M. Epinephrine infusion in the evaluation of unexplained cardiac arrest and familial sudden death: from the cardiac arrest survivors with preserved Ejection Fraction Registry. Circ Arrhythm Electrophysiol. 2012 Oct;5(5):933-40. doi: 10.1161/CIRCEP.112.973230. Epub 2012 Sep 3. PMID 22944906
- [Derived] Krahn AD, Healey JS, Simpson CS, Chauhan VS, Birnie DH, Champagne J, Gardner M, Sanatani S, Chakrabarti S, Yee R, Skanes AC, Leong-Sit P, Ahmad K, Gollob MH, Klein GJ, Gula LJ, Sheldon RS. Sentinel symptoms in patients with unexplained cardiac arrest: from the cardiac arrest survivors with preserved ejection fraction registry (CASPER). J Cardiovasc Electrophysiol. 2012 Jan;23(1):60-6. doi: 10.1111/j.1540-8167.2011.02185.x. Epub 2011 Sep 28. PMID 21955300
- [Derived] Derval N, Simpson CS, Birnie DH, Healey JS, Chauhan V, Champagne J, Gardner M, Sanatani S, Yee R, Skanes AC, Gula LJ, Leong-Sit P, Ahmad K, Gollob MH, Haissaguerre M, Klein GJ, Krahn AD. Prevalence and characteristics of early repolarization in the CASPER registry: cardiac arrest survivors with preserved ejection fraction registry. J Am Coll Cardiol. 2011 Aug 9;58(7):722-8. doi: 10.1016/j.jacc.2011.04.022. PMID 21816308